CLINICAL TRIAL: NCT02130752
Title: Ultrasonic Scalpel vs. Monopolar Electrocautery for D2 Distal Gastric Carcinoma Surgery: a Multicenter Randomized Controlled Trial
Brief Title: Ultrasonic Scalpel vs. Monopolar Electrocautery for D2 Distal Gastric Carcinoma Surgery
Acronym: CGCT-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jian-Kun Hu, Deputy director of Department of Gastrointestinal Surgery, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CGCT-01
Record Dates: First submitted 2014-04-07; First posted 2014-05-05 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer; Surgery; Ultrasonic Scalpel; Monopolar Electrocautery; Operation Time; Blood Loss, Surgical; Quality of Life; External Causes of Morbidity and Mortality
Keywords: Stomach Neoplasms; Operative Time; Gastrectomy; Surgical Hemorrhage; Mortality; Morbidity
MeSH Terms: conditions — Stomach Neoplasms; Blood Loss, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonic scalpel surgery group (Experimental): During the procedures of the abdominal approach D2 distal gastrectomy, use ultrasonic scalpel (Device) to coagulation and cut off blood vessel, separate and dissection lymph-nodes; some great vessels can ligation by nylon, silk line or Hemolock.
  Interventions: Device: Ultrasonic scalpel
- Monopolar electrocautery surgery group (Experimental): During the procedures of the abdominal approach D2 distal gastrectomy, use monopolar electrocautery (Device) to coagulation and cut off blood vessel, separate and dissection lymph-nodes; some great vessels can ligation by nylon, silk line or Hemolock.
  Interventions: Device: Monopolar electrocautery

INTERVENTIONS:
Device: Monopolar electrocautery — During the procedures of the abdominal approach D2 distal gastrectomy, use the monopolar electrocautery (Device) to coagulation and cut off blood vessel, separate and dissection lymph-nodes .
  Arms: Monopolar electrocautery surgery group
Device: Ultrasonic scalpel — During the procedures of the abdominal approach D2 distal gastrectomy, use ultrasonic scalpel (Device) to coagulation and cut off blood vessel, separate and dissection lymph-nodes
  Arms: Ultrasonic scalpel surgery group

SUMMARY:
Gastric cancer as one of the most common gastrointestinal cancers, radical resection of primary lesions combined with dissection of regional lymph-nodes is acknowledged by surgeons all over the world. By the invented and adopted energy surgical instruments, surgical procedure is safer and easier than before. The newly surgical instruments reduce the post-operative mortality and morbidity combined easy procedures of surgery. As the most popular instruments used in the gastric surgery, ultrasonic scalpel and monopolar electrocautery were received lots of attention and concern. Some studies have shown some advantage of the two instruments, which were they can facilitate the surgical treatment and make the surgery safer and more effective. Although, some small retrospective sample reports claimed that ultrasonic scalpel brought benefit in blood loss, dissection lymph-node intraoperative complications and even postoperative complications. And Korea small sample randomized controlled trail presentation that ultrasonic scalpel can reduced blood loss and surgical duration. However, postoperative complications were with no statistical significance between the two instruments. Cost- effective analysis of the energy instruments is still controversial. Large sample randomized control trail with high quality is needed.

By the reasons above, a multicenter randomized controlled trial conducted by 9 hospitals from North to South in China aims to compare the clinical characteristics and outcomes, when using of the ultrasonic scalpel or monopolar electrocautery in traditional open gastrectomy. The aim of this study is to evaluate the outcomes of ultrasonic scalpel compared with monopolar electrocautery in D2 distal gastrectomy, include, intraoperative parameters, postoperative complications, cost data, and post-operative quality of life.

DETAILED DESCRIPTION:
Standard Operating Procedure (SOP)

1. Preoperative evaluation Patients satisfied with inclusion/exclusion criteria will be informed to join in the clinical study and signature the inform consent.
2. Randomization preoperative evaluation found that R0, D2 Gastrectomy can be performed, the case will entrance into the Randomization period. Random numbers are computer-generated, with the third party applications.
3. Surgical procedures The surgical treatments is adopted the traditional open gastrectomy approach and adjuvant D2 lymphadenectomy. The SOP of the surgical treatments are according to the Japanese Gastric Cancer treatments guidelines, 2010, Version 3.
4. Postoperative recovery Postoperative recovery period need to collect those relevant parameters of all the patients. All the relevant parameters had definitely definition in the Case Report Form of this study.
5. Follow-up The follow-up of this study divide into two parts, the postoperative quality of life and tumor characteristics outcomes. The information of the postoperative quality of life is collected by the EuroQol-5 Dimensions (EQ-5D) questionnaire in four postoperative time intervals. The tumor related outcomes included long-term postoperative complications, recurrence type, relapse free survival (months) and the overall survival (months).

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative endoscopy and biopsy confirmed gastric adenocarcinoma, and predictively feasible of traditional open D2 distal gastrectomy;
2. Predictively resectable diseases, of preoperative staging Japanese Gastric Cancer Association (JGCA) 14th Edition cT2N0M0-T4aN3M0, IB-IIIC, except T4b;
3. Age：≤75 years, or ≥18 years;
4. Without serious disease;
5. Patients without previous history of upper abdominal surgery;
6. WHO performance score <2;
7. No limit to sexual and race;
8. informed consent required;

Exclusion Criteria:

1. primary lesion cannot be resected in the pattern of transabdominal distal gastrectomy, but for total gastrectomy, Whipple's procedure, or combined organ resection (include the cholecystectomy) or with a transthoracic approach surgery;
2. Patient undergo emergency surgery due to bleeding or perforation;
3. Patients with other gastric malignant diseases, such as lymphoma and stromal tumors, etc;
4. Patients suffering from malignant diseases before the study;
5. Patients with other severe complications cannot tolerate surgery: such as severe heart and lung diseases, heart function below clinical stage 2, uncontrollable hypertension, pulmonary infection, moderate to severe Chronic Obstruction Pulmonary Disease (COPD), chronic bronchitis, severe diabetes and / or renal insufficiency, severe hepatitis and / or function below the rank of CHILD B grade, and severe malnutrition, etc.
6. Patients treated with neoadjuvant chemotherapy or radiation therapy which might affect the efficacy observation;
7. Severity mental diseases;
8. After signature the Clinical trial agreement, patients and their agent will quit the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Surgical duration | Intraoperative
  From the skin incision to finish the suture of abdominal wall

SECONDARY OUTCOMES:
Blood loss | Intraoperative
  The intraoperative blood loss
Number of harvested and positive lymph nodes | Postoperative
  Number of harvested and positive lymph nodes by pathological results
Intraoperative Mortality and Morbidity | Intraoperative
  Evaluation the intraoperative mortality and morbidity
Survival outcome | 3 years
  the survival outcomes include the 3-year overall survival rate and 3-year disease free survival rate
Postoperative Mortality and Morbidity | Postoperative (30 days)
  Evaluation the postoperative (30 days) mortality and morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Kun Hu, Ph.D., M.D., Principal Investigator — West China Hospital
Locations (9):
- China (9):
  - Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Harbin Medical University, Harbin, Heilongjiang
  - Union Hospital, Tongji Medical College, Wuhan, Hubei
  - The First Affiliated Hospital of China Medical University, Shengyang, Liaoning
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Wu J, Wang H, Yin X, Wang Y, Lu Z, Zhang J, Zhang Y, Xue Y. Normalization weighted combination scores re-evaluate TNM staging of gastric cancer: a retrospective cohort study based on a multicenter database. Int J Surg. 2024 Jan 1;110(1):11-22. doi: 10.1097/JS9.0000000000000726. PMID 38000074